CLINICAL TRIAL: NCT00444028
Title: Safety, Tolerability, and Pharmacokinetics of a Single Dose of Staccato™ Loxapine for Inhalation in Normal, Healthy Volunteers
Brief Title: Staccato Loxapine Single Dose PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMDC-004-101
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2007-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia, Staccato Loxapine
MeSH Terms: conditions — Schizophrenia | interventions — Loxapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort A: Inhaled Loxapine 0.625 mg or Placebo (Experimental): Single 0.625 mg dose of inhaled loxapine or Single Placebo dose of inhaled loxapine
  Interventions: Drug: inhaled Loxapine 0.625 mg; Drug: inhaled Placebo (0 mg)
- Cohort B: Inhaled Loxapine 1.25 mg or Placebo (Experimental): Single 1.25 mg dose of inhaled loxapine or Single Placebo dose of inhaled loxapine
  Interventions: Drug: inhaled Loxapine 1.25 mg; Drug: inhaled Placebo (0 mg)
- Cohort C: Inhaled Loxapine 2.5 mg or Placebo (Experimental): Single 2.5 mg dose of inhaled loxapine or Single Placebo dose of inhaled loxapine
  Interventions: Drug: inhaled Loxapine 2.5 mg; Drug: inhaled Placebo (0 mg)
- Cohort D: Inhaled Loxapine 5 mg or Placebo (Experimental): Single 5 mg dose of inhaled loxapine or Single Placebo dose of inhaled loxapine
  Interventions: Drug: inhaled Loxapine 5 mg; Drug: inhaled Placebo (0 mg)
- Cohort E: Inhaled Loxapine 10 mg or Placebo (Experimental): Single 10 mg dose of inhaled loxapine or Single Placebo dose of inhaled loxapine
  Interventions: Drug: inhaled Loxapine 10 mg; Drug: inhaled Placebo (0 mg)

INTERVENTIONS:
Drug: inhaled Loxapine 0.625 mg — Single 0.625 mg (lowest) dose of inhaled loxapine
  Other Names: ADASUVE
  Arms: Cohort A: Inhaled Loxapine 0.625 mg or Placebo
Drug: inhaled Loxapine 1.25 mg — Single 1.25 mg (2nd) dose of inhaled loxapine
  Other Names: ADASUVE
  Arms: Cohort B: Inhaled Loxapine 1.25 mg or Placebo
Drug: inhaled Loxapine 2.5 mg — Single 2.5 mg (3rd) dose of inhaled loxapine
  Other Names: ADASUVE
  Arms: Cohort C: Inhaled Loxapine 2.5 mg or Placebo
Drug: inhaled Loxapine 5 mg — Single 5 mg (4th) dose of inhaled loxapine
  Other Names: ADASUVE
  Arms: Cohort D: Inhaled Loxapine 5 mg or Placebo
Drug: inhaled Loxapine 10 mg — Single 10 mg (5th) dose of inhaled loxapine
  Other Names: ADASUVE
  Arms: Cohort E: Inhaled Loxapine 10 mg or Placebo
Drug: inhaled Placebo (0 mg) — Single placebo dose of inhaled loxapine
  Other Names: PLACEBO

SUMMARY:
The objective of this study was to assess the safety, tolerability and pharmacokinetics of a single inhaled dose of (administered in 1 or 2 puffs) Staccato Loxapine in healthy volunteers.

DETAILED DESCRIPTION:
Safety and pharmacokinetic data obtained from 50 subjects (between the ages of 18 to 55 years) entered into this randomized, placebo-controlled study. To obtain 50 enrolled subjects, screening procedures and inclusion/exclusion criteria were evaluated for 126 subjects during a variable screening period of up to 21 days. Once enrolled, subjects were randomized to either Staccato Loxapine or Staccato placebo.

Plasma samples for pharmacokinetic analysis were collected beginning on Day 0, pre-dose and continuing for 24 hr post dose. Blood samples for the PK analysis of loxapine and its metabolites (8-OH loxapine, 7-OH loxapine and amoxapine) were obtained at time 0 (immediately before dosing), at 30 sec, 1, 2, 3, 5, 10, 30, 45 min, 1, 2, 4, 6, 12, 24 hr after dosing. Plasma concentrations of loxapine and metabolites were used to estimate the following PK parameters for loxapine and its metabolites: area under the plasma concentration time curve from time 0 extrapolated to infinity (AUCinf), AUC from time 0 to time tlast, the last quantifiable concentration (AUClast), maximum observed plasma concentration (Cmax), observed time of Cmax (tmax), terminal phase elimination rate constant (ke), apparent terminal elimination half life calculated from ke (T½ ), apparent total body clearance / fraction absorbed calculated from AUCinf and dose (CL/F) (for loxapine and the metabolites where permitted by measurable concentrations).

Safety was evaluated by the incidence of adverse events, clinical laboratory testing (blood chemistry, hematology, and urinalysis), physical examination, vital signs, pulse oximetry, postural vital signs, 12-lead electrocardiogram, pulmonary function tests, continuous 12-lead Holter monitoring, sedation assessments, akathisia assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between the ages of 18 to 55 years, inclusive.
2. Subjects with a body mass index (BMI) ≥21 and ≤30.
3. Subjects who speak, read, and understand English and are willing and able to provide written informed consent on an IRB-approved form prior to the initiation of any study procedures.
4. Subjects who are willing and able to be confined to the Clinical Research Unit (CRU) for approximately 2 days and comply with the study schedule and study requirements.
5. Subjects who are in good general health as determined by a complete medical history, physical examination, 12-lead ECG, spirometry, blood chemistry profile, hematology, and urinalysis.

Exclusion Criteria:

1. Subjects who regularly consume large amounts of xanthine-containing substances (i.e., more than 5 cups of coffee or equivalent amounts of xanthine-containing substances per day).
2. Subjects who have taken prescription or nonprescription medication (with the exception of vitamins and acetaminophen if medically necessary) within 5 days of Visit 2 (Baseline).
3. Subjects who have had an acute illness within 5 days of Visit 2 (Baseline).
4. Subjects who have received an investigational drug within 30 days (or within 5 half lives of the investigational drug, if >30 days) prior to Visit 2 (Baseline).
5. Subjects who have smoked tobacco within the last year.
6. Subjects who have a history within the past 2 years of drug or alcohol dependence or abuse as defined by DSM-4.
7. Subjects with a history of HIV positivity.
8. Subjects with a history of allergy or intolerance to dibenzoxazepines (amoxapine and loxapine).
9. Subjects with a known history of contraindications to anticholinergics (bowel obstructions, urinary retention, acute glaucoma).
10. Subjects with a history of pheochromocytoma, seizure disorder, Parkinson's disease, or Restless Leg Syndrome (RLS).
11. Subjects who test positive for alcohol or have a positive urine drug screen at Visit 1 or Visit 2.
12. Subjects who have hypotension (systolic blood pressure ≤90 mmHg, diastolic blood pressure ≤50 mmHg), or hypertension (systolic blood pressure ≥140 mmHg, diastolic blood pressure ≥90 mmHg).
13. Subjects who have a clinically significant ECG abnormality.
14. Subjects with a history of unstable angina, syncope, coronary artery disease, myocardial infarction, congestive heart failure (CHF), stroke, transient ischemic attack (TIA), or a neurological disorder.
15. Subjects who have a history of pulmonary disease that precludes administration of Staccato Loxapine (asthma, bronchitis, bronchospasm, emphysema).
16. Subjects who have an FEV1 less than 80% of predicted values on spirometry assessments at Visit 1.
17. Female subjects who are breastfeeding or have a positive pregnancy test at Visit 1 or Visit 2.
18. Female participants of child-bearing potential or within 1 year of menopause, and sexually active are excluded unless they use a medically acceptable and effective birth control method throughout the study and for 1 week following the end of the study. Medically acceptable methods of contraception include abstinence, diaphragm with spermicide, intrauterine device (IUD), condom with foam or spermicide, vaginal spermicidal suppository, surgical sterilization, and birth control pills. Unacceptable methods include: the rhythm method, withdrawal, condoms alone, or diaphragm alone.
19. Subjects who have any other disease or condition, by history, physical examination, or laboratory abnormalities that in the investigator's opinion, would present undue risk to the subject, or may confound the interpretation of study results.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2005-09; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall Stoltz, MD, Principal Investigator — West Pharmaceutical Services, GFI Research Center, Evansville, IN 47714
Locations (1):
- Covance Clinical Research Unit Inc., d/b/a Covance GFI Research, Evansville, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD submitted to regulatory authorities. Others may contact Alexza Pharmaceuticals, Inc. Please send your request to ClinicalTrialsInfo@alexza.com

REFERENCES:
- [Result] Spyker DA, Munzar P, Cassella JV. Pharmacokinetics of loxapine following inhalation of a thermally generated aerosol in healthy volunteers. J Clin Pharmacol. 2010 Feb;50(2):169-79. doi: 10.1177/0091270009347866. Epub 2009 Nov 13. PMID 19915181

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty subjects were recruited by and studied in the clinical researech unit (CRU). Study dates: 30 September 2005 through 22 November 2005
Pre-assignment Details: To obtain 50 enrolled subjects, screening procedures and inclusion/exclusion criteria were evaluated for 126 subjects during a variable screening period of up to 21 days. No enrolled participants were excluded from the trial.
Groups:
- Placebo: Staccato placebo inhalation device(s)
- Staccato Loxapine 0.625 mg: inhalation of loxapine from a single 0.625 mg device
- Staccato Loxapine 1.25 mg: inhalation of loxapine from a two 0.625 mg devices
- Staccato Loxapine 2.5 mg: inhalation of loxapine from a single 2.5 mg device
- Staccato Loxapine 5 mg: inhalation of loxapine from a single 5 mg device
- Staccato Loxapine 10 mg: inhalation of loxapine from a two 5 mg devices
Period: Overall Study
Arm/Group | Placebo | Staccato Loxapine 0.625 mg | Staccato Loxapine 1.25 mg | Staccato Loxapine 2.5 mg | Staccato Loxapine 5 mg | Staccato Loxapine 10 mg
Started | 14 | 7 | 8 | 6 | 7 | 8
Completed | 14 | 7 | 8 | 6 | 7 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Staccato Loxapine 0.625 mg | Staccato Loxapine 1.25 mg | Staccato Loxapine 2.5 mg | Staccato Loxapine 5 mg | Staccato Loxapine 10 mg | Total
Number analyzed (Participants) | 14 | 7 | 8 | 6 | 7 | 8 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 7 | 8 | 6 | 7 | 8 | 50
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (10.55) | 33.4 (10.44) | 28 (7.11) | 28.2 (6.05) | 30.1 (13.53) | 27.4 (7.65) | 31.7 (10.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 4 | 4 | 5 | 3 | 27
  Male | 6 | 4 | 4 | 2 | 2 | 5 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 7 | 8 | 6 | 7 | 8 | 50

OUTCOME MEASURES:

1. Primary Outcome: Tmax
Description: Tmax = time from inhalation to to maximum observed loxapine concentration
Time Frame: predose, 0.5, 1, 2, 3, 5, 10, 30 and 45 min, 1, 2, 4, 6, 12, and 24 hours
Population: PK Population (N=36) All subjects exposed to inhaled loxapine who provided concentration data
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Staccato Loxapine 0.625 mg | Staccato Loxapine 1.25 mg | Staccato Loxapine 2.5 mg | Staccato Loxapine 5 mg | Staccato Loxapine 10 mg
Number analyzed (Participants) | 7 | 8 | 6 | 7 | 8
minutes | 12.6 (21.3) | 2.15 (1.31) | 2.87 (3.62) | 2.13 (0.687) | 5.25 (10)

2. Primary Outcome: Half-life
Description: Half-life of the terminal elimination phase of loxapine concentrations
Time Frame: predose, 0.5, 1, 2, 3, 5, 10, 30 and 45 min, 1, 2, 4, 6, 12, and 24 hours
Population: PK Population (N=36) All subjects exposed to inhaled loxapine who provided concentration data
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Staccato Loxapine 0.625 mg | Staccato Loxapine 1.25 mg | Staccato Loxapine 2.5 mg | Staccato Loxapine 5 mg | Staccato Loxapine 10 mg
Number analyzed (Participants) | 7 | 8 | 6 | 7 | 8
hours | 5.2 (1.3) | 6.56 (1.44) | 6.92 (1.94) | 6.2 (1.14) | 6.14 (2.16)

3. Primary Outcome: ke
Description: elimination rate constant
Time Frame: predose, 0.5, 1, 2, 3, 5, 10, 30 and 45 min, 1, 2, 4, 6, 12, and 24 hours
Population: PK Population (N=36) All subjects exposed to inhaled loxapine who provided concentration data
Measure: Mean (Standard Error); unit: /hour
Arm/Group | Staccato Loxapine 0.625 mg | Staccato Loxapine 1.25 mg | Staccato Loxapine 2.5 mg | Staccato Loxapine 5 mg | Staccato Loxapine 10 mg
Number analyzed (Participants) | 7 | 8 | 6 | 7 | 8
/hour | .143 (.047) | .111 (.026) | .108 (.033) | .115 (.020) | .122 (.032)

4. Primary Outcome: Clearance
Description: clearance (CL/F) of lozxapine
Time Frame: predose, 0.5, 1, 2, 3, 5, 10, 30 and 45 min, 1, 2, 4, 6, 12, and 24 hours
Population: PK Population (N=36) All subjects exposed to inhaled loxapine who provided concentration data
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Staccato Loxapine 0.625 mg | Staccato Loxapine 1.25 mg | Staccato Loxapine 2.5 mg | Staccato Loxapine 5 mg | Staccato Loxapine 10 mg
Number analyzed (Participants) | 7 | 8 | 6 | 7 | 8
L/hour | 56.2 (14.1) | 55.9 (13.7) | 61.1 (18.8) | 53.8 (9.74) | 78 (25.8)

5. Primary Outcome: Cmax
Description: maximum concentration of loxapine observed
Time Frame: predose, 0.5, 1, 2, 3, 5, 10, 30 and 45 min, 1, 2, 4, 6, 12, and 24 hours
Population: PK Population (N=36) All subjects exposed to inhaled loxapine who provided concentration data
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Staccato Loxapine 0.625 mg | Staccato Loxapine 1.25 mg | Staccato Loxapine 2.5 mg | Staccato Loxapine 5 mg | Staccato Loxapine 10 mg
Number analyzed (Participants) | 7 | 8 | 6 | 7 | 8
ng/mL | 6.5 (8.79) | 9.7 (3.49) | 62.9 (63) | 105 (80.6) | 134 (118.8)

6. Primary Outcome: Dose Proportionality (AUCinf) by Power Analysis
Description: Dose proportionality by power analysis examines the linear regression of the log-AUC versus log-Dose on a by-patient basis across all doses administered. The slope and 90% confidence interval (CI) provide a clear, quantitative (best practices) assessment of the relationship of drug delivered to dose administered. The units on such analyses are generally those of slope (rise over run), with 1.000 being "perfect". Although any positive slope might be considered clinically useful, a 90% CI within the criteria of 0.800-1.250 may be considered a delivery system which is "as good as it gets".
Time Frame: predose, 0.5, 1, 2, 3, 5, 10, 30 and 45 min, 1, 2, 4, 6, 12, and 24 hours
Population: PK Population (N=36) All subjects exposed to inhaled loxapine who provided concentration data
Measure: Mean (Standard Deviation); unit: hr*mcg/L
Arm/Group | Staccato Loxapine 0.625 mg | Staccato Loxapine 1.25 mg | Staccato Loxapine 2.5 mg | Staccato Loxapine 5 mg | Staccato Loxapine 10 mg
Number analyzed (Participants) | 7 | 8 | 6 | 7 | 8
hr*mcg/L | 11.9 (3.70) | 23.4 (4.87) | 44.6 (14.7) | 95.5 (16.6) | 140.6 (44.6)
Statistical Analysis 1: Comparison: Staccato Loxapine 0.625 mg vs Staccato Loxapine 1.25 mg vs Staccato Loxapine 2.5 mg vs Staccato Loxapine 5 mg vs Staccato Loxapine 10 mg; Dose proportionality by power analysis examines the linear regression of the log-AUC versus log-Dose on a by-patient basis across all doses administered. The slope and 90% confidence interval (CI) provide a clear, quantitative (best practices) assessment of the relationship of drug delivered to dose administered; Test type: Other — The units on such analyses are generally those of slope (rise over run), with 1.000 being "perfect". Although any positive slope might be considered clinically useful, a 90% CI within the criteria of 0.800-1.250 may be considered a delivery system which is "as good as it gets"; Slope = 0.909, 90% CI 2-sided [0.832 to 0.987]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were considered treatment related from the first exposure to study treatment until 30 days after the last treatment
Description: Adverse events (AEs) were assessed at 17 pre-specified time points for the 24-hour period after dosing, as well as whenever spontaneously reported by the subjects or study staff
Arm/Group | Placebo | Staccato Loxapine 0.625 mg | Staccato Loxapine 1.25 mg | Staccato Loxapine 2.5 mg | Staccato Loxapine 5 mg | Staccato Loxapine 10 mg
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/7 | 0/8 | 0/6 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/7 | 0/8 | 0/6 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 6/14 | 4/7 | 5/8 | 3/6 | 5/7 | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | Staccato Loxapine 0.625 mg (N=7) | Staccato Loxapine 1.25 mg (N=8) | Staccato Loxapine 2.5 mg (N=6) | Staccato Loxapine 5 mg (N=7) | Staccato Loxapine 10 mg (N=8)
Dysgeusia (Gastrointestinal disorders) | 0 | 1 | 2 | 2 | 2 | 6
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 1 | 1
Fatigue (General disorders) | 1 | 0 | 1 | 1 | 3 | 3
Pallor (General disorders) | 0 | 0 | 0 | 0 | 0 | 3
Disturbance in Attention (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 5 | 2 | 2 | 3 | 4 | 6
Headache (Nervous system disorders) | 2 | 0 | 2 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 3 | 1 | 2 | 0 | 2 | 6

LIMITATIONS AND CAVEATS:
Absolute bioavailability was not determined because loxapine for intravenous comparator was not available comercially in the US

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less